CLINICAL TRIAL: NCT03207815
Title: A Phase 2, Randomized, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Filgotinib in Subjects With Active Noninfectious Uveitis
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in Adults With Active Noninfectious Uveitis
Acronym: HUMBOLDT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-432-4097; 2017-001485-17 (EudraCT Number)
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Noninfectious Uveitis
MeSH Terms: interventions — GLPG0634; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Filgotinib (Experimental): Participants will receive filgotinib 200 milligrams (mg) once daily for up to 52 weeks along with a standardized prednisone burst of 60 milligrams per day (mg/day) at Day 1/Baseline followed by a protocol-defined mandatory taper schedule up to Week 15.
  Interventions: Drug: Filgotinib; Drug: Prednisone
- Placebo (Placebo Comparator): Participants will receive placebo to match filgotinib once daily for up to 52 weeks along with a standardized prednisone burst of 60 mg/day at Day 1/Baseline followed by a protocol-defined mandatory taper schedule up to Week 15.
  Interventions: Drug: Placebo to match filgotinib; Drug: Prednisone

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib
Drug: Placebo to match filgotinib — Tablet(s) administered orally
  Arms: Placebo
Drug: Prednisone — Tablet(s) administered orally

SUMMARY:
The primary objective of this study is to evaluate the efficacy of filgotinib versus placebo for the treatment of the signs and symptoms of noninfectious uveitis as measured by the percentage of participants failing treatment for active noninfectious uveitis by Week 24.

ELIGIBILITY:
Key Inclusion Criteria:

* Is diagnosed with active noninfectious intermediate-, posterior-, or pan-uveitis
* Must have active uveitic disease at the Day 1/Baseline visit as defined by the presence of at least 1 of the following parameters in at least one eye despite 2 weeks of maintenance therapy with oral prednisone (≥ 10 mg/day to ≤ 60 mg/day) or an oral corticosteroid equivalent:

  * Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion
  * ≥ 2+ anterior chamber cells per the Standardization of Uveitis Nomenclature (SUN) criteria
  * ≥ 2+ vitreous haze per the National Eye Institute/Standardization of Uveitis Nomenclature (NEI/SUN) criteria
* No evidence of active tuberculosis (TB) or untreated latent TB

Key Exclusion Criteria:

* Participants with elevated intraocular pressures and/or severe glaucoma
* Confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus (CMV), Human T-Lymphotropic Virus Type 1 (HTLV-1), Whipple's disease, Herpes Zoster virus (HZV), Lyme disease, toxoplasmosis and herpes simplex virus (HSV)

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (24):
- United States (15):
  - Stanford Byers Eye Institute, Palo Alto, California
  - Colorado Retina Associates PC, Golden, Colorado
  - Northwestern Medical Group, Chicago, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - Duke University Eye Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation-Cole Eye Institute, Cleveland, Ohio
  - Oregon Health Science University-Casey Eye Institute, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Texas Retina Associates - Fort Worth, Fort Worth, Texas
  - Foresight Studies, LLC, San Antonio, Texas
  - university of Wisconsin-Madison, Madison, Wisconsin
- Lions Eye Institute, Nedlands, Western Australia, Australia
- Retina Consultants, Vancouver, Canada
- St. Franziskus Hospital, Münster, Germany
- Hadassah Medical Center, Jerusalem, Israel
- Auckland Eye, Remuera, New Zealand
- United Kingdom (4):
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Central Mancester Hospitals NHS Foundation Trust, Manchester Royal Eye Hospital, Manchester
  - Eye Research Group Oxford, Oxford Eye Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava SK, Watkins TR, Nguyen QD, Sharma S, Scales DK, Dacey MS, Shah RE, Chu DS, Grewal DS, Faia LJ, Suhler EB, Genovese MC, Guo Y, Barchuk WT, Besuyen R, Dick AD, Rosenbaum JT. Filgotinib in Active Noninfectious Uveitis: The HUMBOLDT Randomized Clinical Trial. JAMA Ophthalmol. 2024 Sep 1;142(9):789-797. doi: 10.1001/jamaophthalmol.2024.2439. PMID 39023880
- [Derived] Hashida N, Nishida K. Recent advances and future prospects: Current status and challenges of the intraocular injection of drugs for vitreoretinal diseases. Adv Drug Deliv Rev. 2023 Jul;198:114870. doi: 10.1016/j.addr.2023.114870. Epub 2023 May 10. PMID 37172783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, the United Kingdom, Canada, Australia, Germany, Israel, and New Zealand. The first participant was screened on 26 July 2017. The last study visit occurred on 22 April 2021.
Pre-assignment Details: 116 participants were screened.
Groups:
- Filgotinib: Participants received filgotinib 200 milligrams (mg) tablet orally, once daily for up to 52 weeks along with a standardized prednisone burst of 60 mg/day at Day 1/Baseline followed by a protocol-defined mandatory taper schedule up to Week 15.
- Placebo: Participants received placebo to match filgotinib tablet orally, once daily for up to 52 weeks along with a standardized prednisone burst of 60 mg/day at Day 1/Baseline followed by a protocol-defined mandatory taper schedule up to Week 15.
Period: Overall Study
Arm/Group | Filgotinib | Placebo
Started | 38 | 36
Completed | 30 | 29
Not Completed | 8 | 7
Not completed — Protocol Violation | 3 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Investigator's Discretion | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Pregnancy/Partner Pregnancy | 1 | 0
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Filgotinib: Participants received filgotinib 200 mg tablet orally, once daily for up to 52 weeks along with a standardized prednisone burst of 60 mg/day at Day 1/Baseline followed by a protocol-defined mandatory taper schedule up to Week 15.
- Total: Total of all reporting groups
Arm/Group | Filgotinib | Placebo | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15.1) | 43 (15.7) | 46 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 4 | 10 | 14
    Ethnicity: Not Hispanic or Latino | 32 | 25 | 57
    Ethnicity: Not Permitted | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 0 | 4
  Race: Black or African American | 2 | 8 | 10
  Race: Native Hawaiian or Pacific Islander | 1 | 0 | 1
  Race: White | 29 | 26 | 55
  Race: Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
  United Kingdom | 4 | 2 | 6
  Canada | 2 | 0 | 2
  Australia | 1 | 0 | 1
  Germany | 0 | 1 | 1
  Israel | 0 | 1 | 1
  New Zealand | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Failing Treatment for Active NonInfectious Uveitis by Week 24
Description: Treatment failure was a participant meeting at least 1 of these criteria in at least 1 eye: New active, inflammatory lesions relative to Day 1/Baseline (all visits starting Week (Wk) 6); Inability to achieve ≤Grade 0.5+ (at Wk 6) or 2-step increase (change of Grade 0 to Grade 2+/Grade 0.5+ to Grade 3+) (all visits after Wk 6) relative to best state (RBS) achieved in Anterior Chamber (AC) cell grade (Standardization of Uveitis Nomenclature [SUN] criteria)[AC cell grades range from 0 (0 cells) to 4+ (>50 cells), higher scores=severe uveitis]; Inability to achieve ≤Grade 0.5+ (at Wk 6) or 2-step increase (all visits after Wk 6) RBS achieved in Vitreous Haze (VH) grade (National Eye Institute [NEI]/SUN criteria)[VH grades range from 0 (no evident VH) to 4+ (optic nerve head is obscured), higher scores=severe uveitis]; Worsening of best corrected visual acuity (BCVA) by ≥15 letters RBS achieved (all visits starting Wk 6), measured by an eye chart, fewer correct letters=severe uveitis.
Time Frame: Week 6 through Week 24
Population: Evaluable Analysis Set included all randomized participants who received at least one dose of study drug and did not permanently discontinue from the study prior to Week 6.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
percentage of participants | 37.5 [19.2 to 55.8] | 67.6 [50.5 to 84.8]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel — P-value was estimated from the Cochran-Mantel-Haenszel (CMH) test, adjusted for the stratification factors; Participants with missing values on treatment failure status were analyzed as treatment failures using a nonresponder imputation (NRI) method; Difference in Treatment Failure Rate = -30.1, 95% CI 2-sided [-56.2 to -4.1]

2. Secondary Outcome: Time to Treatment Failure on or After Week 6
Description: Treatment failure was a participant meeting at least 1 of these criteria in at least 1 eye: New active, inflammatory lesions relative to Day 1/Baseline (all visits starting Wk 6); Inability to achieve ≤Grade 0.5+ (at Wk 6) or 2-step increase (change of Grade 0 to Grade 2+/Grade 0.5+ to Grade 3+) (all visits after Wk 6) relative to best state (RBS) achieved in AC cell grade (SUN criteria) [AC cell grades range from 0 (0 cells) to 4+ (>50 cells), higher scores=severe uveitis]; Inability to achieve ≤Grade 0.5+ (at Wk 6) or 2-step increase (all visits after Wk 6) RBS achieved in VH grade (NEI/SUN criteria) [VH grades range from 0 (no evident VH) to 4+ (optic nerve head is obscured), higher scores=severe uveitis]; Worsening of BCVA by ≥15 letters RBS achieved (all visits starting Wk 6), measured by an eye chart, fewer correct letters=severe uveitis.
Time Frame: Week 6 through Week 52
Population: Participants in the Evaluable Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
weeks | NA [24.1 to NA] — Not Available as the calculated percentiles of event rate were not reached. | 22.0 [12.1 to 47.0]
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.0014, Stratified Log-Rank Test — P-value was derived from the log rank test stratified by the stratification factors; Stratified Hazard Ratio = 0.309, 95% CI 2-sided [0.144 to 0.663] — Stratified hazard ratio (95% confidence interval [CI]) were derived from the Cox model stratified by the stratification factors

3. Secondary Outcome: Change in Vitreous Haze (VH) Grade in Each Eye (NEI/SUN Criteria), From Best State Achieved Prior to Week 6 to Week 52 or End of Treatment (EOT) Visit or Early Termination (ET)
Description: Grading of VH was based on the publication from the NEI which has also been adapted by the SUN working group. VH grades range from 0 (no evident VH) to 4+ (optic nerve head is obscured), with higher scores indicating greater severity of uveitis. A negative change from best state value obtained prior to Week 6 indicates improvement.
Time Frame: Prior to Week 6; Up to Week 52 or EOT or ET (maximum: 53 weeks)
Population: Participants in the Evaluable Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
score
  Left Eye: Best State Prior to Week 6: number analyzed (Participants) | 32 | 33
  Left Eye: Best State Prior to Week 6 | 0.3 (0.40) | 0.2 (0.33)
  Right Eye: Best State Prior to Week 6 | 0.3 (0.36) | 0.3 (0.45)
  Left Eye: Change From Best State at Week 52/EOT/ET: number analyzed (Participants) | 32 | 33
  Left Eye: Change From Best State at Week 52/EOT/ET | 0.1 (0.79) | 0.3 (0.75)
  Right Eye: Change From Best State at Week 52/EOT/ET: number analyzed (Participants) | 32 | 33
  Right Eye: Change From Best State at Week 52/EOT/ET | 0.1 (0.62) | 0.2 (0.66)
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.3550, Repeated Measure ANCOVA — P-value was estimated using a repeated measure Analysis of Covariance (ANCOVA) model which included treatment, eye, interaction of treatment and eye, stratification factors and best state value; The repeated measure ANCOVA model was used to control for the clustered observations from each eye of a participant; Least Squares Mean Treatment Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14 — Treatment difference in Least Squares (LS)-means (95% CI) were obtained from the repeated measure ANCOVA model

4. Secondary Outcome: Change in Anterior Chamber (AC) Cell Grade in Each Eye, From Best State Achieved Prior to Week 6 to Week 52 or EOT Visit or ET
Description: The number of AC cells observed within a 1 mm × 1 mm slit beam were recorded for each eye. The reported number was used to determine the grade according to the SUN criteria. AC cell grades range from 0 (0 cells in field) to 4+ (>50 cells in field), with higher scores indicating more cells visible in the AC and greater severity of uveitis. A negative change from best state value obtained prior to Week 6 indicates improvement.
Time Frame: Prior to Week 6; Up to Week 52 or EOT or ET (maximum: 53 weeks)
Population: Participants in the Evaluable Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
score
  Left Eye: Best State Prior to Week 6 | 0.0 (0.09) | 0.1 (0.19)
  Right Eye: Best State Prior to Week 6 | 0.0 (0.12) | 0.1 (0.25)
  Left Eye: Change From Best State at Week 52/EOT/ET | 0.2 (0.59) | 0.6 (0.87)
  Right Eye: Change From Best State at Week 52/EOT/ET | 0.2 (0.53) | 0.7 (1.05)
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.0145, Repeated Measure ANCOVA — P-value was estimated using a repeated measure ANCOVA model which included treatment, eye, interaction of treatment and eye, stratification factors and best state value; The repeated measure ANCOVA model was used to control for the clustered observations from each eye of a participant; LS Mean Treatment Difference = -0.4, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.18 — Treatment difference in LS-means (95% CI) were obtained from the repeated measure ANCOVA model

5. Secondary Outcome: Change in Logarithm of the Minimal Angle of Resolution (logMAR) Best Corrected Visual Acuity (BCVA) in Each Eye, From Best State Achieved Prior to Week 6 to Week 52 or EOT Visit or ET
Description: BCVA is the best possible vision that an eye can achieve with the set of glasses or contact lenses. A refraction test was performed to measure the appropriate lens strength to focus light on the retina. Using the appropriate corrective lenses based on that visit's refraction, participant's BCVA was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. In the ETDRS system, 15 letters is equal to a change in 3 lines of visual acuity. If the participant is unable to read letters on a testing chart, visual acuity is described as ranging from ability to count fingers, recognize hand movements, or light perception. The smaller BVCA score indicates greater severity of uveitis. A positive change from best state value obtained prior to Week 6 indicates improvement.
Time Frame: Prior to Week 6; Up to Week 52 or EOT or ET (maximum: 53 weeks)
Population: Participants in the Evaluable Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
logMAR
  Left Eye: Best State Prior to Week 6 | 0.09 (0.195) | 0.07 (0.209)
  Right Eye: Best State Prior to Week 6 | 0.09 (0.193) | 0.12 (0.280)
  Left Eye: Change From Best State at Week 52/EOT/ET | 0.03 (0.154) | 0.05 (0.112)
  Right Eye: Change From Best State at Week 52/EOT/ET | -0.01 (0.116) | 0.07 (0.144)
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.0389, Repeated Measure ANCOVA — [p-value comment as in outcome 4, analysis 1]; The repeated measure ANCOVA model was used to control for the clustered observations from each eye of a participant; LS Mean Treatment Difference = -0.05, 95% CI 2-sided [-0.10 to -0.00], Standard Error of Mean 0.025 — Treatment difference in LS-means (95% CI) were obtained from the repeated measure ANCOVA model

6. Secondary Outcome: Log Change in Central Retinal Thickness in Each Eye, From Best State Achieved Prior to Week 6 to Week 52 or EOT Visit or ET
Description: Central retinal thickness is measured by optical coherence tomography (OCT). Central retinal thickness is defined as the thickness of the retina in the center of the foveal pit (1 mm subfield). The larger central retinal thickness value indicates greater severity of uveitis. A negative change from best state value obtained prior to Week 6 indicates improvement.
Time Frame: Prior to Week 6; Up to Week 52 or EOT or ET (maximum: 53 weeks)
Population: Participants in the Evaluable Analysis Set with the available data were analyzed.
Measure: Mean (Standard Deviation); unit: log microns
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
log microns
  Left Eye: Best State Prior to Week 6 | 2.45 (0.059) | 2.46 (0.097)
  Right Eye: Best State Prior to Week 6 | 2.47 (0.056) | 2.44 (0.104)
  Left Eye: Change From Best State at Week 52/EOT/ET: number analyzed (Participants) | 32 | 32
  Left Eye: Change From Best State at Week 52/EOT/ET | 0.01 (0.062) | 0.04 (0.080)
  Right Eye: Change From Best State at Week 52/EOT/ET: number analyzed (Participants) | 32 | 32
  Right Eye: Change From Best State at Week 52/EOT/ET | 0.01 (0.049) | 0.03 (0.055)
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.0340, Repeated Measure ANCOVA — P-value was estimated using a repeated measure ANCOVA model which included treatment, eye, interaction of treatment and eye, OCT machine, and best state value; The repeated measure ANCOVA model was used to control for the clustered observations from each eye of a participant; LS Mean Treatment Difference = -0.02, 95% CI 2-sided [-0.05 to -0.00], Standard Error of Mean 0.011 — Treatment difference in LS-means (95% CI) were obtained from the repeated measure ANCOVA model

7. Secondary Outcome: Time to Development of Macular Edema in At Least One Eye on or After Week 6
Description: Time in weeks until the development of Macular edema or Week 52 or EOT or ET. Macular edema is determined by OCT and is defined as central retinal thickness ≥ 300 microns if using Cirrus machine, or ≥ 315 microns if using Spectralis machine.
Time Frame: Week 6 through Week 52
Population: Participants in the Evaluable Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Filgotinib | Placebo
Number analyzed (Participants) | 32 | 34
weeks | 7.8 [6.1 to NA] — Not Available as the calculated percentiles of event rate were not reached. | 12.3 [6.1 to NA] — Not Available as the calculated percentiles of event rate were not reached.
Statistical Analysis 1: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.5893, Stratified Log-Rank Test — P-value was derived from the log rank test stratified by the stratification factors; Stratified Hazard Ratio = 1.193, 95% CI 2-sided [0.625 to 2.277] — Stratified hazard ratio (95% CI) were derived from the Cox model stratified by the stratification factors

8. Secondary Outcome: Plasma Concentration of Filgotinib
Time Frame: Day 1 post dose, Weeks 4 and 6 predose, Week 12 post dose, Weeks 24, 36, 52 (EOT), ET at any time
Population: Participants in the Safety Analysis Set who have at least one non-missing concentration data with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/ml)
Arm/Group | Filgotinib
Number analyzed (Participants) | 37
nanograms per millilitre (ng/ml)
  Day 1 Postdose | 748.5 (1043.84)
  Week 4 Predose: number analyzed (Participants) | 29
  Week 4 Predose | 173.3 (364.46)
  Week 6 Predose: number analyzed (Participants) | 28
  Week 6 Predose | 133.9 (306.18)
  Week 12 Postdose: number analyzed (Participants) | 27
  Week 12 Postdose | 1088.7 (856.57)
  Week 24 Single Anytime: number analyzed (Participants) | 21
  Week 24 Single Anytime | 397.5 (561.57)
  Week 36 Single Anytime: number analyzed (Participants) | 14
  Week 36 Single Anytime | 295.7 (420.25)
  Week 52 Single Anytime: number analyzed (Participants) | 22
  Week 52 Single Anytime | 195.2 (344.54)
  Early Termination Single Anytime: number analyzed (Participants) | 3
  Early Termination Single Anytime | 434.8 (478.72)

9. Secondary Outcome: Plasma Concentration of Metabolite, GS-829845
Time Frame: Day 1 post dose, Weeks 4 and 6 predose, Week 12 post dose, Weeks 24, 36, 52 (EOT), ET at any time
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Filgotinib
Number analyzed (Participants) | 37
ng/ml
  Day 1 Postdose | 230.8 (317.98)
  Week 4 Predose: number analyzed (Participants) | 29
  Week 4 Predose | 2085.6 (924.91)
  Week 6 Predose: number analyzed (Participants) | 28
  Week 6 Predose | 2107.7 (749.28)
  Week 12 Postdose: number analyzed (Participants) | 27
  Week 12 Postdose | 3237.0 (1180.74)
  Week 24 Single Anytime: number analyzed (Participants) | 21
  Week 24 Single Anytime | 3478.1 (1137.63)
  Week 36 Single Anytime: number analyzed (Participants) | 14
  Week 36 Single Anytime | 2944.3 (1130.84)
  Week 52 Single Anytime: number analyzed (Participants) | 22
  Week 52 Single Anytime | 2510.7 (1732.59)
  Early Termination Single Anytime: number analyzed (Participants) | 3
  Early Termination Single Anytime | 2171.0 (1224.77)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 30 days after the last dose of study drug (maximum exposure up to 57 weeks); All-Cause Mortality: From randomization up to 57 weeks
Description: Adverse Events: Safety Analysis Set included all participants who received at least 1 dose of study drug.
  All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
Arm/Group | Filgotinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 5/37 | 2/35
Other Adverse Events (participants affected / at risk) | 28/37 | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib (N=37) | Placebo (N=35)
Retinal vasculitis (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib (N=37) | Placebo (N=35)
Anterior chamber inflammation (Eye disorders) | 1 | 2
Cataract (Eye disorders) | 2 | 1
Chalazion (Eye disorders) | 0 | 2
Chorioretinal disorder (Eye disorders) | 2 | 2
Dry eye (Eye disorders) | 2 | 4
Eye irritation (Eye disorders) | 2 | 2
Eye pain (Eye disorders) | 2 | 1
Macular oedema (Eye disorders) | 2 | 1
Ocular hyperaemia (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 2 | 0
Photopsia (Eye disorders) | 3 | 0
Uveitis (Eye disorders) | 2 | 2
Visual impairment (Eye disorders) | 5 | 1
Vitreous floaters (Eye disorders) | 3 | 1
Vitreous haze (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 3 | 3
Bronchitis (Infections and infestations) | 1 | 2
Covid-19 (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 4 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0
Intraocular pressure increased (Investigations) | 2 | 2
Weight increased (Investigations) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 7
Anxiety (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 4 | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypertension (Vascular disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Study was terminated early due to termination of the development program. Due to early termination and small sample size, pharmacokinetic (PK) analysis was not performed for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03207815/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT03207815/SAP_001.pdf